CLINICAL TRIAL: NCT03225937
Title: Open-Label, Phase II Study of Trastuzumab in Combination With Lapatinib (Cohort A) or Pertuzumab in Combination With Trastuzumab-emtansine (Cohort B) in Patients With HER2-positive Metastatic Colorectal Cancer: the HERACLES (HER2 Amplification for Colo-rectaL Cancer Enhanced Stratification)Trial
Brief Title: Evaluation of Trastuzumab in Combination With Lapatinib or Pertuzumab in Combination With Trastuzumab-Emtansine to Treat Patients With HER2-positive Metastatic Colorectal Cancer
Acronym: HERACLES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 004-IRCC-10IIS-12; 2012-002128-33 (EudraCT Number)
Record Dates: First submitted 2017-06-13; First posted 2017-07-21 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trastuzumab; Lapatinib; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: two sequential cohorts: cohort A (lapatinib + trastuzumab); cohort B (pertuzumab + trastuzumab-emtansine).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Trastuzumab and lapatinib
  Interventions: Drug: Trastuzumab, Lapatinib
- Cohort B (Experimental): Pertuzumab and Trastuzumab-emtansine
  Interventions: Drug: Pertuzumab, trastuzumab-emtansine

INTERVENTIONS:
Drug: Trastuzumab, Lapatinib — Patients enrolled in Cohort A will receive lapatinib 1000 mg daily per os + trastuzumab 4 mg/kg iv load, followed by 2 mg/kg iv weekly. Patients will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever come first.
  Arms: Cohort A
Drug: Pertuzumab, trastuzumab-emtansine — Patients enrolled in Cohort B will receive pertuzumab 840 mg iv load, followed by 420 mg iv Q3weeks + trastuzumab-emtansine 3.6 mg/kg iv on day 1 of each subsequent 3 week cycle.
  Patients will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever come first.
  Arms: Cohort B

SUMMARY:
This is a Phase II multi-center 2-sequential cohorts trial, designed to assess the objective response rate of two anti HER2 combination in advanced disease CRC patients harbouring an amplified HER2 tumor assessed according to HERACLES Diagnostic Criteria by FISH/SISH.

Cohort A: monoclonal antibody trastuzumab, used in combination with the small molecule tyrosine kinase inhibitor lapatinib.

Cohort B, monoclonal antibody pertuzumab, used in combination with the antibody drug conjugate trastuzumab-emtansine.

Please note that cohort A accrual has been closed and endpoint already reached.

DETAILED DESCRIPTION:
Investigators identified HER2 amplification as a potential onco-driver and marker of de novo resistance to anti-EGFR therapy in mCRC patients for which other known genetic alterations conferring resistance to anti EGFR antibodies were excluded.

Exploiting direct transfer xenografts of mCRC surgical samples in mice (xenopatients), investigators conducted a multi-arm study in HER2-amplified xenopatients showing that combinations of the dual EGFR/HER2 inhibitor lapatinib and the anti-HER2 moAb trastuzumab induced long-lasting tumor regressions, while monotherapy with lapatinib led to stabilization and monotherapy with trastuzumab was ineffective. On these findings investigators designed the HERACLES trial.

HERACLES is an open-label Phase II, 2-sequential cohorts trial, assessing the response rate (ORR) of Trastuzumab combined Lapatinib (Cohort A) or Pertuzumab combined with trastuzumab-emtansine (Cohort B), in metastatic colorectal patients harboring an amplified HER2 tumors .

HER2 positivity is centrally established by immunohistochemistry (IHC) and Silver In Situ Hybridization (SISH). To be HER2 eligible the original tumor, or the biopsied metastasis (whichever is last available), must be IHC 3+ or 2+ in more than 50% of cells, confirmed by SISH or FISH with a HER2:CEP17 ratio ≥ 2.0. For IHC a positive staining (3+) is defined as an intense membrane staining which can be circumferential, basolateral, or lateral of the tumor cells.

ELIGIBILITY:
Inclusion criteria COHORT A

1. Histological/confirmed adenocarcinoma of the colon or rectum with metastatic disease not amenable to salvage surgery.
2. Pathology mandatory requirements: the original tumour specimen must be KRAS WT and SISH/FISH positive or IHC 3+ positive in more than 50% cells. Note: for immunohistochemistry a positive staining (3+) is defined as an intense membrane staining which can be circumferential, basolateral, or lateral of the tumor cells. the original paraffin block or a minimum of 15 polarized unstained slides from the original paraffin block must be made available to the Pathology Core within 15 days from registration.
3. Age ≥18
4. ECOG PS 0-1
5. Measurable disease as defined by RECIST 1.1 criteria.
6. Progression (PD) while on, or within 6 months from therapy with approved standard drugs.
7. Unless otherwise contraindicated patients should have received and failed the following previous therapies for mCRC: fluoropyrimidines, oxaliplatin, irinotecan, cetuximab or panitumumab containing regimens. Bevacizumab is allowed
8. Adequate haematological function as defined by: ANC > 1.5 x 109/L, platelet count >100 x 109/L, haemoglobin > 10 g/dL
9. Adequate renal function, as defined by: creatinine < 1.5 x UNL
10. Adequate hepatobiliary function, as defined by the following baseline liver function tests: total serum bilirubin <1.5 upper normal limit (UNL); alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 2.5xUNL; alkaline phosphatase (AP) < 2.5xUNL, if total alkaline phosphatase (AP) > 2.5xUNL, alkaline phosphatase liver fraction must be < 2.5xUNL
11. Adequate contraception for all fertile patients
12. Negative pregnancy test

Exclusion criteria COHORT A

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Radiotherapy ≤ 4 weeks prior to enrolment.
2. Other chemotherapy or biological therapy treatment ≤ 4 weeks prior to enrolment.
3. Symptomatic brain metastases.
4. Active infection.
5. Gastro-intestinal abnormalities, inability to take oral medication, any condition affecting absorption.
6. Impaired cardiac function including any of the following: uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; chronic heart failure (CHF) of New York Heart Association (NYHA) Grade II or higher (See Appendix 4); or serious cardiac arrhythmia requiring medication, baseline Left Ventricular Ejection Fraction (LVEF) ≤ 55% measured by echocardiography (ECHO).
7. Major surgery in the two weeks prior to entering the clinical trial.
8. Concurrent treatment with any other anti-cancer therapy.
9. History of another neoplastic disease (except basal cell carcinoma of the skin or uterine cervix carcinoma in situ adequately treated), unless in remission for ≥ 5 years.
10. Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
11. Pregnant and lactating women.
12. Patients with history of hypersensitivity to either IP or excipients.
13. Men and women of childbearing potential who are not using an effective method of contraception.
14. Participation in another clinical trial or treatment with any investigational product within 4 weeks prior to inclusion in this study.
15. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
16. Patient with unresolved hypokalaemia, hypomagnesemia or hypocalcaemia

Inclusion criteria COHORT B

1. Histological/confirmed adenocarcinoma of the colon or rectum with metastatic disease not amenable to salvage surgery.
2. The original tumour specimen must be RAS (KRAS exons 2 3 4; NRAS exons 2 3 4) wild type and SISH/FISH positive or IHC 2+/3+ positive in more than 50% cells.
3. Age ≥18.
4. ECOG PS 0-1.
5. Measurable disease as defined by RECIST 1.1 criteria.
6. Progression (PD) while on, or within 6 months from therapy with approved standard drugs.
7. Unless otherwise contraindicated, patients must have received and failed fluoropyrimidines, oxaliplatin, irinotecan -containing regimens as previous therapies for metastatic disease.
8. Patients having failed only one line of chemotherapy for their metastatic diseases are eligible if they have received:
9. FOLFOXIRI;
10. FOLFIRI after progression to adjuvant FOLFOX, occurred on treatment or within 6 months after treatment completion.
11. Treatments with bevacizumab, aflibercept or regorafenib and cetuximab or panitumumab are allowed.
12. Adequate hematological function as defined by: ANC <= 1.5 x 109/L, platelet count >=100 x 109/L, haemoglobin >= 10 g/dL
13. Adequate renal function, as defined by: creatinine <= 1.5 x UNL
14. Adequate hepato-biliary function, as defined by the following baseline liver function tests:

    1. total serum bilirubin <=1.5 upper normal limit (UNL)
    2. alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 2.5xUNL
    3. alkaline phosphatase (AP) <= 2.5xUNL; if total alkaline phosphatase (AP) > 2.5xUNL, alkaline phosphatase liver fraction must be <= 2.5xUNL
15. Adequate contraception for all fertile patients
16. Negative pregnancy test

Exclusion criteria COHORT B

1. Radiotherapy <= 4 weeks prior to enrolment.
2. Other chemotherapy or biological therapy treatment ≤ 4 weeks prior to enrolment.
3. Symptomatic brain metastases.
4. Active infection.
5. Gastro-intestinal abnormalities, inability to take oral medication, any condition affecting absorption.
6. Impaired cardiac function including any of the following: uncontrolled hypertension (systolic >150 mmHg and/or diastolic > 100 mmHg) or clinically significant (ie active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication; unstable angina; chronic heart failure (CHF) of New York Heart Association (NYHA) Grade II or higher (See Appendix 4); or serious cardiac arrhythmia requiring medication, baseline Left Ventricular Ejection Fraction (LVEF) ≤ 55% measured by echocardiography (ECHO).
7. Major surgery in the two weeks prior to entering the clinical trial.
8. Concurrent treatment with any other anti-cancer therapy.
9. History of another neoplastic disease (except basal cell carcinoma of the skin or uterine cervix carcinoma in situ adequately treated), unless in remission for ≥ 5 years
10. Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.
11. Pregnant and lactating women.
12. Patients with history of hypersensitivity to either IP or excipients.
13. Men and women of childbearing potential who are not using an effective method of contraception.
14. Participation in another clinical trial or treatment with any investigational product within 4 weeks prior to inclusion in this study.
15. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
16. Patient with unresolved hypokalaemia, hypomagnesemia or hypocalcaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate according to RECIST 1.1 criteria | Time Frame: every 8 weeks (cohort A) or every 9 weeks (cohort B) from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months

SECONDARY OUTCOMES:
Description of the frequency and severity of Adverse Events based on the NCI -CTCAE V4.0 | Time Frame: weekly (cohort A) or every 21 days (cohort B) from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
Progression Free Survival | Time Frame: every 8 weeks (cohort A) or every 9 weeks (cohort B) from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Siena, MD, Study Chair — Grande Ospedale Metropolitano Niguarda - Milano
Locations (7):
- Italy (7):
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, Please Select
  - AOU Policlinico S. Orsola Malpighi, Bologna
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Seconda Università di Napoli, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Campus Biomedico, Roma
  - AOU Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valtorta E, Martino C, Sartore-Bianchi A, Penaullt-Llorca F, Viale G, Risio M, Rugge M, Grigioni W, Bencardino K, Lonardi S, Zagonel V, Leone F, Noe J, Ciardiello F, Pinto C, Labianca R, Mosconi S, Graiff C, Aprile G, Frau B, Garufi C, Loupakis F, Racca P, Tonini G, Lauricella C, Veronese S, Truini M, Siena S, Marsoni S, Gambacorta M. Assessment of a HER2 scoring system for colorectal cancer: results from a validation study. Mod Pathol. 2015 Nov;28(11):1481-91. doi: 10.1038/modpathol.2015.98. Epub 2015 Oct 9. PMID 26449765
- [Result] Sartore-Bianchi A, Trusolino L, Martino C, Bencardino K, Lonardi S, Bergamo F, Zagonel V, Leone F, Depetris I, Martinelli E, Troiani T, Ciardiello F, Racca P, Bertotti A, Siravegna G, Torri V, Amatu A, Ghezzi S, Marrapese G, Palmeri L, Valtorta E, Cassingena A, Lauricella C, Vanzulli A, Regge D, Veronese S, Comoglio PM, Bardelli A, Marsoni S, Siena S. Dual-targeted therapy with trastuzumab and lapatinib in treatment-refractory, KRAS codon 12/13 wild-type, HER2-positive metastatic colorectal cancer (HERACLES): a proof-of-concept, multicentre, open-label, phase 2 trial. Lancet Oncol. 2016 Jun;17(6):738-746. doi: 10.1016/S1470-2045(16)00150-9. Epub 2016 Apr 20. PMID 27108243
- [Derived] Sartore-Bianchi A, Lonardi S, Martino C, Fenocchio E, Tosi F, Ghezzi S, Leone F, Bergamo F, Zagonel V, Ciardiello F, Ardizzoni A, Amatu A, Bencardino K, Valtorta E, Grassi E, Torri V, Bonoldi E, Sapino A, Vanzulli A, Regge D, Cappello G, Bardelli A, Trusolino L, Marsoni S, Siena S. Pertuzumab and trastuzumab emtansine in patients with HER2-amplified metastatic colorectal cancer: the phase II HERACLES-B trial. ESMO Open. 2020 Sep;5(5):e000911. doi: 10.1136/esmoopen-2020-000911. PMID 32988996